CLINICAL TRIAL: NCT00345293
Title: A Phase I/II Study of Autologous Dendritic Cells Pulsed With Apoptotic Tumor Cells (DC/PC3) Administered Subcutaneously to Prostate Cancer Patients.
Brief Title: Dendritic Cell Vaccine Study (DC/PC3) for Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDA-0537
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC/PC3 vaccine (Experimental): 3 subcutaneous injections of ex vivo-generated autologous dendritic cell vaccine: 1) pulsed with apoptotic PC3 cells; 2) pulsed with apoptotic PC3-M1 cells, and 3) pulsed with keyhole limpet hemocyanin (KLH, control antigen)
  Interventions: Biological: autologous dendritic cell vaccine (DC/PC3)

INTERVENTIONS:
Biological: autologous dendritic cell vaccine (DC/PC3) — ex vivo generated autologous dendritic cells pulsed with apoptotic PC3 cells and pulsed with apoptotic PC3-M1 cells(control apoptotic cells) and pulsed with KLH (control antigen). maximum dose of DC/PC3 that we are able to generate from their initial leukaphereses product, up to a maximum of 10 x 106 DCs. Doses in the range of 105 to 10 x 106 DCs have been used clinically without toxicity

SUMMARY:
The purpose of this study is to assess the safety and activity of DC/PC3, a dendritic cell vaccine used as immunotherapy for prostate cancer. The vaccine is made with each participants' own immune cells obtained through blood donation. Dendritic cells are known to activate other immune cells such as T cells, that are able to mount an attack against cancer cells. The dendritic cell vaccine will be administered as injections every 2 weeks over a course of 2 months.

DETAILED DESCRIPTION:
See Brief Summary.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer

Rising prostate specific antigen (PSA, 3 values, each measured at least 2 weeks apart) post initial therapy (ie, radiation, prostatectomy) human leukocyte antigen A2.1 (HLA-A2.1)

-

Exclusion Criteria:

central nervous system metastasis

History of autoimmune disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-06; Primary Completion 2013-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Darnell, MD PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Frank MO, Kaufman J, Parveen S, Blachere NE, Orange DE, Darnell RB. Dendritic cell vaccines containing lymphocytes produce improved immunogenicity in patients with cancer. J Transl Med. 2014 Dec 5;12:338. doi: 10.1186/s12967-014-0338-3. PMID 25475068
- See also: study description at Rockefeller University website — http://clinicalstudies.rucares.org/protocol.php?id=262&cat=50&sub=5

RESULTS

PARTICIPANT FLOW:
Groups:
- DC/PC3 Vaccine-selected: 3 subcutaneous injections of ex vivo-generated autologous dendritic cell vaccine: 1) autologous dendritic cell vaccine (DC/PC3): ex vivo generated autologous dendritic cells pulsed with apoptotic PC3 cells and 2) pulsed with apoptotic PC3-M1 cells (control apoptotic cells) and 3) pulsed with KLH (control antigen). Maximum dose of DC/PC3 that we are able to generate from their initial leukaphereses product, up to a maximum of 10 x 10^6 DCs. DCs were made from precursors isolated using antibodies.
- DC/PC3- Adherent: 3 subcutaneous injections of ex vivo-generated autologous dendritic cell vaccine: 1) autologous dendritic cell vaccine (DC/PC3): ex vivo generated autologous dendritic cells pulsed with apoptotic PC3 cells and 2) pulsed with apoptotic PC3-M1 cells (control apoptotic cells) and 3) pulsed with KLH (control antigen). Maximum dose of DC/PC3 that we are able to generate from their initial leukaphereses product, up to a maximum of 10 x 10^6 DCs. DCs were made from precursors isolated using the adherence method.
Period: Overall Study
Arm/Group | DC/PC3 Vaccine-selected | DC/PC3- Adherent
Started | 10 | 3
Completed | 8 | 3
Not Completed | 2 | 0
Not completed — Unable to access line for sample | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | DC/PC3 Vaccine
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 64 [53 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: adverse events
Time Frame: through week 29
Measure: Number; unit: events
Arm/Group | DC/PC3 Vaccine
Number analyzed (Participants) | 13
events
  Serious Adverse Events | 2
  Other Adverse Events | 204

2. Secondary Outcome: Immunogenicity
Description: The Tritiated thymidine proliferation assay is used to assess samples collected pre-treatment and those collected post-treatment; the outcome measure is the change in counts per minute (post-treatment counts minus pre-treatment counts).
Time Frame: pre and post treatment
Population: One other participant in DC/PC3 vaccine-Selected group not analyzed due to failed controls in assay.
Measure: Median (Full Range); unit: counts per minute
Groups:
- DC/PC3 Vaccine- Selected: 3 subcutaneous injections of ex vivo-generated autologous dendritic cell vaccine: 1) pulsed with apoptotic PC3 cells; 2) pulsed with apoptotic PC3-M1 cells, and 3) pulsed with keyhole limpet hemocyanin (KLH, control antigen)
  autologous dendritic cell vaccine (DC/PC3): ex vivo generated autologous dendritic cells pulsed with apoptotic PC3 cells and pulsed with apoptotic PC3-M1 cells (control apoptotic cells) and pulsed with KLH (control antigen).
  Dendritic cells were made from antibody selected cells.
- DC/PC3- Adherent: 3 subcutaneous injections of ex vivo-generated autologous dendritic cell vaccine: 1) pulsed with apoptotic PC3 cells; 2) pulsed with apoptotic PC3-M1 cells, and 3) pulsed with keyhole limpet hemocyanin (KLH, control antigen)
  autologous dendritic cell vaccine (DC/PC3): ex vivo generated autologous dendritic cells pulsed with apoptotic PC3 cells and pulsed with apoptotic PC3-M1 cells (control apoptotic cells) and pulsed with KLH (control antigen).
  Dendritic cells were made from the adherent subset of peripheral blood mononuclear cells.
Arm/Group | DC/PC3 Vaccine- Selected | DC/PC3- Adherent
Number analyzed (Participants) | 7 | 3
counts per minute | 62 [-112 to 4493] | 9461 [985 to 9985]

3. Secondary Outcome: Clinical Response
Time Frame: Post treatment
Population: This data was not collected due to differences in immunogenicity based on different dendritic cell preparations. This data was no longer relevant.
Arm/Group | DC/PC3 Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Common toxicity criteria v4
Arm/Group | DC/PC3 Vaccine
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DC/PC3 Vaccine (N=13)
chest pain (Cardiac disorders) | 1 (1)
arrhythmia (Cardiac disorders) | 1 (1) — hospitalization for pacemaker placement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DC/PC3 Vaccine (N=13)
absolute lymphocyte, low (Blood and lymphatic system disorders) | 1 (1) — G1
acid phosphatase, high (General disorders) | 1 (1) — G1
albumin, low (Blood and lymphatic system disorders) | 1 (1) — G1
albumin, trace, urine (General disorders) | 2 (3) — G1
alkaline phosphatase, high (General disorders) | 1 (1) — G1
ALT, high (Gastrointestinal disorders) | 1 (1) — G2
ANA, high (General disorders) | 2 (2) — G1
ANC, low (Blood and lymphatic system disorders) | 1 (1) — G2
AST, high (Hepatobiliary disorders) | 2 (2) — G1 and G3
bacteria, urine, few (General disorders) | 1 (1) — G1
basophil, high (Blood and lymphatic system disorders) | 1 (1) — G1
bilirubin, urine, small (General disorders) | 1 (1) — G1
blood, urine, trace (Renal and urinary disorders) | 2 (3) — G1
BUN, high (General disorders) | 1 (3) — G1
calcium, ionized, low (General disorders) | 1 (1) — G1
chloride, high (General disorders) | 4 (6) — G1
CO2, high (General disorders) | 7 (12) — G1
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — G1
creatinine, high (Blood and lymphatic system disorders) | 3 (4) — G1 and G2
crystals, urine (Renal and urinary disorders) | 2 (2) — G1
diarrhea (Gastrointestinal disorders) | 1 (1) — G1
fatigue (General disorders) | 2 (5) — G1 and G2
glucose, high (General disorders) | 3 (4) — G1 and G2
glucose, low (General disorders) | 2 (3) — G1 and G2
headache (General disorders) | 1 (1) — G1
heartburn (Gastrointestinal disorders) | 2 (2) — G1 and G2
hematocrit, low (Blood and lymphatic system disorders) | 3 (5) — G1
hematoma (General disorders) | 1 (1) — G1
hemoglobin, low (Blood and lymphatic system disorders) | 2 (2) — G1
hemorrhage, GU, bladder (Renal and urinary disorders) | 1 (2) — G1 and G2
epistaxis (General disorders) | 1 (1) — G1
injection site reaction (General disorders) | 11 (28) — G1 and G2
INR, low (General disorders) | 1 (1) — G1
ketones, urine, high (General disorders) | 2 (3) — G1
leuko est, urine, high (General disorders) | 2 (3) — G1
lightheadedness (General disorders) | 1 (1) — G1
low back pain (General disorders) | 2 (2) — G1
LUC, high (General disorders) | 1 (1) — G1
lymphocytes, %, low (General disorders) | 3 (3) — G1
MCHC, high (Blood and lymphatic system disorders) | 6 (9) — G1
monocytes, %, high (Blood and lymphatic system disorders) | 2 (2) — G1
neutrophils, %, high (Blood and lymphatic system disorders) | 3 (3) — G1
neutrophils, %, low (Blood and lymphatic system disorders) | 1 (1) — G1
numbness/tingling (General disorders) | 2 (2) — G1
chest pain (Cardiac disorders) | 1 (1) — G3
pain (General disorders) | 6 (6) — G1
pH, urine, high (General disorders) | 3 (5) — G1
platelet, high (General disorders) | 1 (1)
platelets, low (General disorders) | 1 (3)
potassium, high (General disorders) | 2 (5) — G1
presyncope (General disorders) | 1 (1) — G2
Prolonged QTc interval (Cardiac disorders) | 1 (1) — G2
pulmonary nodules (General disorders) | 1 (1)
rash (General disorders) | 2 (3) — G1
RBC, low (Blood and lymphatic system disorders) | 3 (5) — G1
RBC, urine, high (Renal and urinary disorders) | 6 (10) — G1
RDW, high (General disorders) | 1 (1)
rheumatoid factor, positive (General disorders) | 1 (1) — G1
rosecea (Skin and subcutaneous tissue disorders) | 1 (1) — G1
seasonal allergies (Immune system disorders) | 1 (1) — G1
specific gravity, urine, high (Renal and urinary disorders) | 5 (6)
specific gravity, urine, low (Renal and urinary disorders) | 4 (5) — G1
swollen glands (General disorders) | 1 (1) — G1
thyroid nodules (General disorders) | 1 (1)
total bilirubin, high (General disorders) | 2 (2)
total protein, low (General disorders) | 1 (2) — G1
URI (General disorders) | 1 (1) — G1
vasovagal episode (General disorders) | 1 (1) — G2
vomiting (Gastrointestinal disorders) | 1 (1)
WBC, low (Blood and lymphatic system disorders) | 3 (4) — G1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes